CLINICAL TRIAL: NCT01725984
Title: AMS AdVance and AdVance XP Male Sling Systems for the Treatment of Stress Urinary Incontinence Following Prostatectomy: Evaluation of Safety, Efficacy, and Quality of Life Through Retrospective Chart Review and Prospective Follow-up
Status: Completed | Type: Observational
Sponsor: American Medical Systems (Industry)
Responsible Party: Sponsor
Other Study IDs: MC1201
Record Dates: First submitted 2012-07-13; First posted 2012-11-14 (Estimated); Results first posted 2015-06-30 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Urinary Incontinence, Stress; Intrinsic Sphincter Deficiency
Keywords: Male Incontinence; AdVance Male Sling; AdVance XP Male Sling; Male Sling
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- AdVance: Subjects previously implanted with the AdVance Male Sling
- AdVance XP: Subjects previously implanted with the AdVance XP male sling

SUMMARY:
A single-center retrospective chart review of AdVance and AdVance XP subject data, combined with prospective follow-up of the same subjects to confirm continence, adverse event, and quality of life status. This study includes patients previously implanted with an AdVance or AdVance XP male sling.

DETAILED DESCRIPTION:
A single-center retrospective chart review of AdVance and AdVance XP subject data, combined with prospective follow-up of the same subjects to confirm continence, adverse event, and quality of life status. This study includes patients previously implanted with an AdVance or AdVance XP male sling.

ELIGIBILITY:
Inclusion Criteria:

1. Valid, written informed consent has been obtained
2. Male subject ≥40 years of age who received the AdVance male sling after January 1, 2010 or the AdVance XP male sling after July 1, 2010 for the treatment of post prostatectomy SUI
3. Pad use of 1 to 8 pads per day prior to sling placement (subjects who used only a dry prophylactic pad or safety liner at baseline will not be included)
4. External (distal) sphincter contractility and a coaptive zone of ≥ 1cm confirmed by endoscopic view prior to sling placement
5. Primary etiology of SUI resulting from radical prostatectomy including, simple open prostatectomy, robotic or laparoscopic prostatectomy

Exclusion Criteria:

1. Pad use of more than 8 pads per day prior to sling placement for incontinence management
2. Urine loss while lying in bed prior to sling placement
3. Treatment with a urethral sling system, an AMS Sphincter 800®, or any implanted device for the treatment of urinary incontinence (not including bulking agents) prior to sling placement
4. TURP procedure prior to sling placement
5. Urge predominant incontinence prior to sling placement
6. Past or current neurological disorder (e.g. neurogenic bladder, multiple sclerosis, Parkinson's disease)
7. History of connective tissue or autoimmune conditions
8. Past or current condition of compromised immune system
9. Placement of an inflatable penile prosthesis (IPP) after sling placement
10. Post void residual of >50 ml prior to sling placement

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male subject ≥40 years of age who received the AdVance male sling after January 1, 2010 or the AdVance XP male sling after July 1, 2010 for the treatment of post prostatectomy SUI at one institution in Munich, Germany.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricarda Bauer, MD, Principal Investigator — Ludwig-Maximilians Universität (LMU)
Locations (1):
- Ludwig-Maximilians Universität (LMU), Munich, Bavaria, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 140 subjects were screened for inclusion into the study. 80 total subjects met all inclusion and none of the exclusion criteria.
Period: Overall Study
Arm/Group | AdVance | AdVance XP
Started | 39 | 41
Completed | 39 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AdVance | AdVance XP | Total
Number analyzed (Participants) | 39 | 41 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.2 (4.9) | 68.8 (5.3) | 69.5 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 39 | 41 | 80
Region of Enrollment [Number; unit: participants]
  Germany | 39 | 41 | 80

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With a ≥50% Reduction in Pads Per Day Use
Description: Evaluate the proportion of subjects with a ≥50% reduction in pads per day use
Time Frame: 3 Months Post Procedure
Measure: Number; unit: percentage of participants
Arm/Group | AdVance | AdVance XP
Number analyzed (Participants) | 39 | 41
percentage of participants | 87.2 | 97.6

2. Primary Outcome: Percentage of Subjects Cured, Improved, or Failed Based on Reported Pad Per Day Use
Description: Evaluate the proportion of subjects cured (0 pads per day or 1 dry prophylactic pad), improved (not cured and ≥50% reduction in pad use), or failed (not cured and not improved) at the three month and final prospective follow-up visit
Time Frame: 3 months Post Procedure
Measure: Number; unit: percentage of subjects
Arm/Group | AdVance | AdVance XP
Number analyzed (Participants) | 39 | 41
percentage of subjects
  Cured | 79.5 | 82.9
  Improved | 7.7 | 14.6
  Failed | 12.8 | 2.4

3. Primary Outcome: Percentage of Subjects in Each Pre-defined Range of Pads Per Day Use
Description: Evaluate the proportion of subjects using the following categories of pads per day at the three month and final prospective follow-up visit:
  0 pads per day or 1 dry prophylactic pad; 1 pad per day; 2 pads per day; 3 pads per day; 4 pads per day; 5 or more pads per day (5, 6, 7, 8 etc. pads per day);
Time Frame: Baseline
Measure: Number; unit: percentage of subjects
Arm/Group | AdVance | AdVance XP
Number analyzed (Participants) | 39 | 41
percentage of subjects
  0 Pads per Day | 0 | 0
  1 Pad per Day | 20.5 | 4.9
  2 Pads per Day | 15.4 | 26.8
  3 Pads per Day | 20.5 | 24.4
  4 Pads per Day | 12.8 | 7.3
  5 or more Pads per Day | 30.8 | 36.6

4. Primary Outcome: Evaluate the 24-hour Pad Weight at the Final Prospective Follow-up Visit
Description: Percentage of subjects at a given weight for their 24-hour pad weight test at the final prospective follow-up visit.
Time Frame: Prospective follow-up to 36 Months Post Procedure
Measure: Number; unit: percentage of subjects
Arm/Group | AdVance | AdVance XP
Number analyzed (Participants) | 39 | 41
percentage of subjects
  <= 10g | 59.0 | 68.3
  10g - 50g | 30.8 | 22.0
  > 50g | 10.3 | 9.8

5. Primary Outcome: Change in Quality of Life Scores as Compared to Baseline for I-QOL, ICIQ-SF, and Summary of Values for the PGI-I. Measured From Baseline to Prospective Follow.
Description: The Incontinence Quality of Life Questionnaire (I-QOL) is a 22 questionnaire that evaluates a subject's quality of life with respect to urinary problems/incontinence. A lower score correlates with more severe incontinence, and an increase from baseline indicates an improvement in quality of life. The score scale is 0 - 100.
  The International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) is a 4 question tool that quantifies the impact on quality of life from incontinence. A decrease from baseline to follow-up indicates an improvement in quality of life. The score scale is 1-21.
  The Patient Global Impression of Improvement (PGI-I) questionnaire is a single question instrument that assess a subject's perception of the disease impact on their quality of life. Completed at the last visit, a lower score indicates a better perception from the patient. Scale from 1 to 7.
Time Frame: Baseline to Prospective Follow Up (up to 36 months)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | AdVance | AdVance XP
Number analyzed (Participants) | 39 | 41
Score on a scale
  IQOL Baseline | 46.5 (21.0) | 45.6 (16.1)
  IQOL 3 Month FU | 81.4 (21.5) | 85.4 (17.8)
  IQOL Prospective FU | 79.9 (21.7) | 86.8 (17.4)
  ICIQ-SF Baseline | 14.4 (5.1) | 15.9 (3.5)
  ICIQ-SF 3 Month FU | 6.1 (5.4) | 4.1 (4.3)
  ICIQ-SF Prospective FU | 6.9 (5.6) | 5.2 (4.6)
  PGI-I Prospective FU | 1.7 (1.1) | 1.4 (1.1)

6. Primary Outcome: Number of Adverse Events Reported Between Arms
Description: Evaluate the occurrence of all AdVance /AdVance XP AEs, as well as those reported as serious, intra-operative, device or procedure related adverse events
Time Frame: Prospective follow-up to 36 Months Post Procedure
Measure: Number; unit: Adverse Events
Arm/Group | AdVance | AdVance XP
Number analyzed (Participants) | 39 | 41
Adverse Events
  Total Number of AEs | 9 | 12
  Procedure Related AEs | 8 | 8
  Device Related AEs | 5 | 8
  Intra-operative | 0 | 0
  Serious | 2 | 3

7. Primary Outcome: Percentage of Subjects With a ≥50% Reduction in Pads Per Day Use
Description: Evaluate the proportion of subjects with a ≥50% reduction in pads per day use
Time Frame: Prospective follow-up to 36 Months Post Procedure
Measure: Number; unit: percentage of subjects
Arm/Group | AdVance | AdVance XP
Number analyzed (Participants) | 39 | 41
percentage of subjects | 69.2 | 90.2

8. Primary Outcome: Percentage of Subjects Cured, Improved, or Failed Based on Reported Pad Per Day Use
Description: as for outcome 2
Time Frame: Prospective follow-up to 36 Months Post Procedure
Measure: Number; unit: percentage of subjects
Arm/Group | AdVance | AdVance XP
Number analyzed (Participants) | 39 | 41
percentage of subjects
  Cured | 46.2 | 65.9
  Improved | 23.1 | 24.4
  Failed | 30.8 | 9.8

9. Primary Outcome: Percentage of Subjects in Each Pre-defined Range of Pads Per Day Use
Description: as for outcome 3
Time Frame: 3 Months Post Procedure
Measure: Number; unit: percentage of subjects
Arm/Group | AdVance | AdVance XP
Number analyzed (Participants) | 31 | 38
percentage of subjects
  0 Pads per Day | 87.1 | 86.8
  1 Pad per Day | 9.7 | 10.5
  2 Pads per Day | 3.2 | 2.6
  3 Pads per Day | 0 | 0
  4 Pads per Day | 0 | 0
  5 Pads per Day | 0 | 0

10. Primary Outcome: Percentage of Subjects in Each Pre-defined Range of Pads Per Day Use
Description: as for outcome 3
Time Frame: Prospective follow-up to 36 Months Post Procedure
Measure: Number; unit: percentage of subjects
Arm/Group | AdVance | AdVance XP
Number analyzed (Participants) | 39 | 41
percentage of subjects
  0 Pads per Day | 46.2 | 65.9
  1 Pad per Day | 23.1 | 12.2
  2 Pads per Day | 10.3 | 17.1
  3 Pads per Day | 12.8 | 0
  4 Pads per Day | 2.6 | 4.9
  5 or more Pads per Day | 5.1 | 0

ADVERSE EVENTS:
Time Frame: All adverse events were collected during the study conductance between August 2012 and January 2013 (6 Months), and were reported from subjects between January 2010 to January 2013 (3 years).
Groups:
- AdVance: Subjects implanted with the AdVance Male Sling
- AdVance XP: Subjects implanted with the AdVance XP Male Sling
Arm/Group | AdVance | AdVance XP
Serious Adverse Events (participants affected / at risk) | 2/39 | 3/41
Other Adverse Events (participants affected / at risk) | 6/39 | 7/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AdVance (N=39) | AdVance XP (N=41)
Infection (Infections and infestations) | 1 (1) | 0
Pain/Discomfort (Surgical and medical procedures) | 1 (1) | 0
Incontinence De Novo (Urge) (Renal and urinary disorders) | 0 | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AdVance (N=39) | AdVance XP (N=41)
Elevated Post-Void Residual (PVR) (Renal and urinary disorders) | 1 (1) | 3 (3)
Superficial Wound Infection (Renal and urinary disorders) | 1 (1) | 0
Urinary Incontinence- De Novo (Stress) (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary Incontinence- De Novo (Urge) (Renal and urinary disorders) | 1 (1) | 0
Urinary Incontinence- Worsening Urge (Renal and urinary disorders) | 0 | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary Urgency (Renal and urinary disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No